CLINICAL TRIAL: NCT00893841
Title: A Randomized, Double-Blind, Placebo Controlled Exploratory Study of Augmentation of Seroquel XR With Pramipexole Dihydrochloride for Bipolar Depression
Brief Title: Bipolar Study of Seroquel XR With Pramipexole Dihydrochloride
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. D McIntosh & Dr. K Kjernisted Clinical Research Inc. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1443C00032
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Bipolar Depression
Keywords: bipolar; bipolar depression; bipolar disorder; depression; quetiapine; pramipexole; Seroquel XR; Mirapex
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Quetiapine Fumarate; Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Quetiapine XR 300mg + Placebo
  Interventions: Drug: quetiapine (Seroquel) XR; Drug: placebo
- 2 (Experimental): Quetiapine XR 300mg + Pramipexole 0.25mg
  Interventions: Drug: quetiapine (Seroquel) XR; Drug: pramipexole dihydrochloride
- 3 (Experimental): Quetiapine XR 300mg + Pramipexole 0.50mg
  Interventions: Drug: quetiapine (Seroquel) XR; Drug: pramipexole dihydrochloride

INTERVENTIONS:
Drug: quetiapine (Seroquel) XR — tablets and caplets, take with liquid before bedtime
  Other Names: Seroquel XR
  Arms: 2; 3
Drug: quetiapine (Seroquel) XR — tablets, take with liquid before bedtime
  Other Names: Seroquel XR
  Arms: 1
Drug: placebo — placebo
  Arms: 1
Drug: pramipexole dihydrochloride — tablets and caplets, take with liquid before bedtime
  Other Names: mirapex
  Arms: 2; 3

SUMMARY:
This study is designed to assess the use of pramipexole dihydrochloride and quetiapine (Seroquel) XR as combination therapy for bipolar depression. The proposed benefit of the combination therapy investigated in this study is improved treatment of bipolar depression.

DETAILED DESCRIPTION:
Quetiapine is a first-line option in Canadian guidelines for the treatment of bipolar depression; however, there is room for improvement as the remission rate is approximately 50% and the response rate is approximately 60%. Pramipexole, which is currently used to treat Parkinson's disease and restless legs syndrome, is reported to have antidepressant effects in patients with unipolar or bipolar depression. There are no other clinical studies to evaluate the efficacy of pramipexole combined with an atypical antipsychotic, such as quetiapine XR, in the treatment of bipolar depression.

This study is a multicentre, randomized, double-blind and placebo-controlled exploratory study in which patients will receive one of three treatment arms for a treatment period of 16 weeks: quetiapine XR plus placebo, quetiapine XR plus 0.25mg pramipexole, or quetiapine XR plus 0.50mg pramipexole.

ELIGIBILITY:
Inclusion Criteria:

* You must be between 18 years and 65 years of age.
* You must have been diagnosed with bipolar depression.
* You must (for women who are able to become pregnant) have a negative urine human chorionic gonadotropin (HCG) pregnancy test at enrolment and be using a reliable form of birth control for the entire duration of the study. The study staff will inform about what is considered an acceptable method of birth control.
* You must provide consent.
* You must be able to understand and comply with the requirements of the study

Exclusion Criteria:

* You are pregnant or lactating (breast-feeding),
* Your symptoms are due to the direct physiological effects of a substance (e.g. drug of abuse, medication, or other treatment) or a general medical condition,
* You have a primary psychotic disorder (e.g., schizophrenia),
* You have a personality disorder diagnosis which in the study doctor's opinion is the focus of clinical concern.
* You have a history or presence of any psychotic illness, including major depression with psychotic features.
* In the opinion of the study doctor, you pose an imminent risk of suicide or a danger to yourself or others,
* You have known allergies to quetiapine or to components of the medication capsule,
* You use any "prohibited" medications. You must inform the study coordinator or study doctor of all the medications that you are taking, and he/she will tell you if any of those medications exclude you from the study.
* You have a substance dependence (drug or alcohol dependence) which in the study doctor's opinion is the focus of clinical concern,
* You have a medical condition that would affect absorption, distribution, metabolism, or excretion of the medication,
* You have an unstable or inadequately treated medical illness (e.g. unstable diabetes, angina pectoris, hypertension) as judged by the study doctor,
* You have diabetes mellitus (DM) which, in the opinion of the study doctor, would exclude you from the study,
* You have an absolute neutrophil count (ANC) of ≤1.5 x 109 per liter
* You are involved in the planning and conduct of the study ,
* You were previously enrolled or randomized in this present study,
* You participated in another drug trial within 4 weeks prior enrolment into this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) total score | Week 0 to Week 16

SECONDARY OUTCOMES:
The mean change in MADRS total score | Week 0 to Week 8
Proportion of subjects achieving remission (MADRS score of less than or equal to 10) | Week 16
Proportion of subjects achieving response (reduction of at least 50% in MADRS total score) | Week 0 to Week 16
Mean change in HAM-D 21 total score | Week 0 to Week 16
Proportion of subjects achieving remission (HAM-D 21 total score of less than or equal to 7) | Week 16
Proportion of subjects achieving treatment response (reduction of at least 50% in HAM-D 21 total score) | Week 0 to Week 16
Mean change in Vancouver Semi-Structured Interview for Depression (V-SID) total score | Week 0 to Week 16
Proportion of subjects withdrawing from study due to inadequate control of depressive symptoms | Week 0 - 16
Change in neurocognitive function, assessed by CNS Vital Signs | Week 0 to Week 16
Change in neuroimmune biological markers | Week 0 to Week 16
Adverse events and patient withdrawal due to adverse events | Week 0 - Week 16
Treatment emergent mania | Week 0 - Week 16
Treatment-emergent extra-pyramidal symptoms | Week 0 - Week 16
Metabolic effects | Week 0 - Week 16

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - Affiliated Research Institute, San Diego, California
  - Eastside Therapeutic Resource, Kirkland, Washington
- Canada (7):
  - Dr. P. Chokka, Edmonton, Alberta
  - Penticton Regional, Penticton, British Columbia
  - Copeman Neuroscience Centre, Vancouver, British Columbia
  - AK Munshi Medical Inc., Sydney, Nova Scotia
  - Regional Mental Health Care - London, London, Ontario
  - Hôpital Louis-H.Lafontaine, Montreal, Quebec
  - Clinique Marie Fitzbach, Québec, Quebec